CLINICAL TRIAL: NCT01889589
Title: Baseline 24 Hour Urine Collection in Population-based Sample of NYC Adults
Brief Title: NYC Heart Follow-Up Study 2010
Acronym: HFUS
Status: Completed | Type: Observational
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Stella Yi, Data & Analytics Group Leader, New York City Department of Health and Mental Hygiene
Other Study IDs: NYCHFUS2010
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Sodium

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- NYC adults
  Interventions: Other: Surveillance

INTERVENTIONS:
Other: Surveillance

SUMMARY:
This surveillance project will assess NYC population sodium intake using the gold standard measurement of 24-hour urine collection. This surveillance project is a critical component of a larger initiative, coordinated by NYC, to reduce sodium intake nationwide through voluntary industry reductions in processed food sodium content. The project will assess current population sodium intake, against which population intake changes at three years can be assessed

ELIGIBILITY:
Inclusion Criteria:

* > 18 Years

Exclusion Criteria:

* Pregnant, breastfeeding or lactating; past or current dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NYC adult population
Sampling Method: Probability Sample
Enrollment: 1775 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
24-hour urinary sodium | 24-hour period

CONTACTS AND LOCATIONS:
Locations (1):
- New York, New York, United States

REFERENCES:
- [Derived] Elfassy T, Yi SS, Llabre MM, Schneiderman N, Gellman M, Florez H, Prado G, Zeki Al Hazzouri A. Neighbourhood socioeconomic status and cross-sectional associations with obesity and urinary biomarkers of diet among New York City adults: the heart follow-up study. BMJ Open. 2017 Dec 29;7(12):e018566. doi: 10.1136/bmjopen-2017-018566. PMID 29289939
- [Derived] Loftfield E, Yi S, Curtis CJ, Bartley K, Kansagra SM. Potassium and fruit and vegetable intakes in relation to social determinants and access to produce in New York City. Am J Clin Nutr. 2013 Nov;98(5):1282-8. doi: 10.3945/ajcn.113.059204. Epub 2013 Sep 11. PMID 24025631